CLINICAL TRIAL: NCT02879929
Title: Development and Validity of the DyNaChron Questionnaire for Chronic Nasal Dysfunction
Acronym: DyNaChron
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GUILLEMIN Francis, MD, PU-PH, Central Hospital, Nancy, France
Other Study IDs: DyNaChron
Record Dates: First submitted 2016-08-19; First posted 2016-08-26 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Rhinitis; Nasal Polyps
Keywords: chronic nasal dysfunction; Quality of life; measurement; self-reporting questionnaire; development; validation
MeSH Terms: conditions — Rhinitis; Nasal Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Nasal symptoms are the main elements that lead to a therapeutic decision and allow for evaluating treatment effects or natural evolution. Despite availability of several questionnaires with good measurement qualities, no systematic assessment takes into account the specific physical and psychosocial consequences of each of the six main nasal symptoms, independently of the disease. The study proposed to measure these symptoms with the use of a selfreport questionnaire and to test the validity of the questionnaire in a large representative sample of patients attending outpatient rhinologic clinics.

DETAILED DESCRIPTION:
The study was conducted in two parts: (1) expert-based development and testing of the face validity of a questionnaire in French; and (2) validity testing, including construct validity by factor analysis, reproducibility by intraclass correlation coefficient (ICC) and Bland and Altman plots, and sensitivity to change by standardized response means, on a large sample of patients in a prospective multicenter study. DyNaChron, a questionnaire with 78 items divided into six domains and exploring both the physical and psychosocial repercussions of CND, was developed. In total, 759 patients completed the questionnaire at a first visit to a clinic, and 539 again 19.5 days later, on average.

ELIGIBILITY:
Inclusion Criteria:Patients had to

* be older than 18 years
* have nasal or sinus dysfunction for more than 3 months
* be able to understand and read theFrench language.

Exclusion Criteria:

* nasal or sinus tumor or Rendu-Osler disease,
* patients were under immediate post-operative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were consecutively recruited in 16 centers in rhinology outpatient clinics all over France.
Sampling Method: Non-Probability Sample
Enrollment: 759 (Actual)
Dates: Start 2005-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Development of the DyNaChron questionnaire for chronic nasal dysfunction | 6 months
  to develop a self-report questionnaire to assess nose and sinus functional symptoms together with their consequences for physical and psychosocial areas

SECONDARY OUTCOMES:
Validation of the DyNaChron questionnaire for chronic nasal dysfunction | 10 months
  to test the validity of the new instrument developped in a large representative sample of patients attending outpatient rhinology clinics

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kacha S, Guillemin F, Jankowski R. Development and validity of the DyNaChron questionnaire for chronic nasal dysfunction. Eur Arch Otorhinolaryngol. 2012 Jan;269(1):143-53. doi: 10.1007/s00405-011-1690-z. Epub 2011 Jul 8. PMID 21739093